CLINICAL TRIAL: NCT02837991
Title: A Phase l Open-Label, Dose Escalation and Cohort Expansion Study, to Assess the Safety and Activity of the Antibody-Drug Conjugate CDX-014 in Advanced or Metastatic Renal Cell Carcinoma (RCC) and Advanced or Metastatic Ovarian Clear Cell Carcinoma (OCCC)
Brief Title: A Dose Escalation, Safety and Activity Study of CDX-014 in Patients With Renal Cell Carcinoma and Ovarian Clear Cell Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development of CDX-014 discontinued
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX014-01
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2018-11

CONDITIONS: Renal Cell Carcinoma (RCC); Clear-cell Renal Cell Carcinoma; Papillary Renal Cell Carcinoma; Kidney Neoplasms; Metastatic Renal Cell Carcinoma; Ovarian Clear Cell Carcinoma
Keywords: Kidney Cancer; Celldex; Dose Escalation; Ovarian Cancer; Ovarian Carcinoma; Kidney Diseases
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Ovarian Neoplasms; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CDX-014 (Experimental): During the treatment phase of the study, patients will receive CDX-014 treatment every 3 weeks (RCC or OCCC) or every 2 weeks (RCC) as long as they remain eligible. Patients may be discontinued from CDX-014 treatment based on the results of disease assessments or if experiencing side effects that make study therapy intolerable.
  The planned dose of CDX-014 depends on the cohort assigned at enrollment.
  Interventions: Drug: CDX-014

INTERVENTIONS:
Drug: CDX-014

SUMMARY:
This is a study to determine the safety of CDX-014 and effectiveness (how well the drug works).

DETAILED DESCRIPTION:
CDX-014 is an antibody-drug conjugate that binds to a protein called TIM-1, which is found on a high percentage of kidney cells that are clear or papillary and ovarian cancer cells that are clear cell.

The study will enroll patients with advanced or metastatic renal cell carcinoma and ovarian clear cell carcinoma to determine the safety and efficacy of CDX-014.

This study will include a Dose-Escalation Phase followed by a Cohort Expansion Phase

All patients enrolled in the study will be closely monitored to determine if there is a response to the treatment as well as for any side effects that may occur.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of advanced or metastatic clear cell or papillary renal cell carcinoma or histologically confirmed clear cell ovarian carcinoma.
2. For RCC, at least two prior anticancer regimens (one must be a VEGF-targeted TKI), or are otherwise inappropriate candidates for all approved therapies. For OCCC, at least one line of prior therapy with a platinum and taxane regimen.
3. Documented progressive disease based on radiographic, clinical or pathologic assessment during or subsequent to last therapy.
4. Measureable (target) disease.
5. Must have available tumor tissue for TIM-1 expression testing
6. Life expectancy ≥ 3 months
7. If of childbearing potential (male or female), agrees to use effective contraception during study treatment and for at least 6 months following last treatment dose.

Exclusion Criteria:

1. Prior therapy containing MMAE
2. Any prior cytotoxic chemotherapy regimen, including antibody drug conjugates for RCC or cytotoxic chemotherapy within 3 weeks of study treatment for OCCC
3. Tyrosine kinase inhibitor (TKI) therapy within 2 weeks or at least 5 half-lives (whichever is longer) prior to planned start of study treatment.
4. Monoclonal antibody therapy within 4 weeks prior to the planned start of study treatment.
5. Radiation therapy within 4 weeks prior to start of study treatment (palliative radiotherapy to bone lesions allowed up to 2 weeks prior to study treatment start).
6. Major surgery or significant traumatic injury within 4 weeks prior to study entry.
7. Use of other investigational drugs within 2 weeks or 5 half-lives (whichever is longer) prior to study treatment.
8. Concurrent severe and/or uncontrolled medical conditions (uncontrolled diabetes or infection), known infection with HIV, Hepatitis B or Hepatitis C.
9. Brain metastases, unless previously treated and asymptomatic and not progressive for 2 months.
10. Significant cardiovascular disease (including congestive heart failure).
11. Other malignancy except for treated and cured basal or squamous cell skin cancer, cured in situ cancers, or other cancer from which the patient has been disease-free for ≥ 3 years.
12. Active systemic infection requiring treatment. Infection controlled by oral therapy will not be exclusionary.
13. Chronic use of systemic corticosteroid above an accepted physiologic dose (5mg per day of prednisone or equivalent) within 7 days of enrollment except when used as premedication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06; Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Dose Escalation - Determine Maximum Tolerated Dose (MTD) | Within 21 days after first dose.
  Determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) of CDX-014 (in mg/kg). MTD will be defined as the highest dose-level where DLT (dose-limiting toxicity) occurs in less than 33% of treated patients.
Cohort Expansion - Assess Objective Response Rate (ORR) | Evaluated every 6-9 weeks following treatment initiation until treatment is discontinued or disease progression, up to 5 years.
  Objective Response Rate (ORR) defined as the proportion of patients who achieve radiographic partial or complete response according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guideline.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Result] McGregor BA, Gordon M, Flippot R, Agarwal N, George S, Quinn DI, Rogalski M, Hawthorne T, Keler T, Choueiri TK. Safety and efficacy of CDX-014, an antibody-drug conjugate directed against T cell immunoglobulin mucin-1 in advanced renal cell carcinoma. Invest New Drugs. 2020 Dec;38(6):1807-1814. doi: 10.1007/s10637-020-00945-y. Epub 2020 May 29. PMID 32472319